CLINICAL TRIAL: NCT03730896
Title: Effectiveness of Dry Needling of the Sternocleidomastoid in Patients With Cervicogenic Headaches - A Randomized Clinical Trial
Brief Title: Effectiveness of Dry Needling of the Sternocleidomastoid in Patients With Cervicogenic Headaches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough viable subjects
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FGCU IRB 2018-49
Record Dates: First submitted 2018-10-29; First posted 2018-11-05 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cervicogenic Headache
Keywords: Dry needling; Cervicogenic headache; Manual therapy
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Masking Description: Random assignment to dry needle group or control group with standard manual therapy interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care group (No Intervention): Normal manual therapy interventions Clinician will decide normal course of treatment
- Dry needling (Experimental): Dryneedling group Clinician will decide normal course of treatment and dry needling of the Sternocleidomastoid muscle (SCM) muscle will be added to that treatment
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Dryneedling of the sternocleidomastoid muscles within a standard treatment approach of physical therapy
  Arms: Dry needling

SUMMARY:
Evaluating the benefit of dry needling of the sternocleidomastoid muscle in subjects with cervicogenic headaches.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether individuals with cervicogenic headache respond favorably to a program of manual therapy in combination with dry needling of the major muscle between chest bone and the head (sternocleidomastoid muscle) compared to manual therapy directed to the upper body quadrant alone.

The researchers will conduct a randomized clinical trial to assess the effectiveness of a manual therapy and dry needling approach (group 1) vs. manual therapy only. (group 2)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years old
2. Primary complaint of cervicogenic headache
3. Restricted cervical Range of motion
4. Neck Disability Index > 20 points

Exclusion Criteria:

1. Red flags identified during the patients physical therapy initial evaluation (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, symptoms of vertebrobasilary insufficiency, pregnancy, cervical spinal stenosis, bilateral upper extremity symptoms etc.
2. Use of blood thinners
3. History of whiplash injury within the past six weeks
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   1. Muscle weakness involving a major muscle group of the upper extremity
   2. Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps)
   3. Diminished or absent sensation to pinprick in any upper extremity dermatome
6. Prior surgery to the neck or thoracic spine
7. Chiropractic, Physical Therapy, or Acupuncture treatment for their neck pain in the last 6-months
8. Workers compensation or pending legal action regarding their headaches
9. Insufficient English language skills to complete all questionnaires
10. Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Headache Disability Index (HDI) score | At initial evaluation (day 1), week three (day 21) and week 6 (day 42)
  Questionnaire for self report, this will be on a 0-100 score

SECONDARY OUTCOMES:
Change in cervical range of motion using an inclinometer/ change in high cervical range of motion using the Flexion-Rotation Test (FRT) | At initial evaluation (day 1), week three (day 21) and week 6 (day 42)
  range of motion assessment, this will be measured in degrees with standardized goniometer measure
Change in the neck disability Index score | At initial evaluation (day 1), week three (day 21) and week 6 (day 42)
  Self report neck pain questionnaire, This is a 0-100 score
Change in visual analogue scale score | At initial evaluation (day 1), week three (day 21) and week 6 (day 42)
  Pain intensity scale,on a 10 cm line patient is asked to mark pain with one vertical mark

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, PhD, Principal Investigator — FGCU Assistent Professor
Locations (1):
- Integrated therapy Practice PC, Hobart, Indiana, United States

IPD SHARING:
Plan to Share IPD: No